CLINICAL TRIAL: NCT01690806
Title: Dexamethasone for the Prevention of Recurrent Laryngeal Nerve Palsy (and Not Only) After Thyroid Surgery. A Randomized Double-blind Placebo-controlled Trial.
Brief Title: Dexamethasone for the Prevention of Recurrent Laryngeal Nerve Palsy
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Aquila (Other)
Responsible Party: Principal Investigator, CECILIA Emanuela Marina, M.D., Università degli Studi dell'Aquila
Other Study IDs: OTO: OTO12-0447R
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2011-08

CONDITIONS: Benign Neoplasm of Thyroid Gland; Malignant Neoplasm of Thyroid
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- dexamethasone: Patients who receive dexamethasone (8 mg; Decadron; Merck Sharp & Dohme) intravenously 90 min before skin incision
- placebo: Patients who receive saline placebo intravenously 90 min before skin incision

SUMMARY:
Recurrent laryngeal nerve dysfunction and hypoparathyroidism are well-recognized important complications of thyroid surgery. The duration of convalescence, after non complicated thyroid operation, may depend on several factors of which pain and fatigue are the most important. Nausea and vomiting occur mainly on the day of operation. Glucocorticoids are well known for their analgesic, anti-inflammatory, immune modulating and antiemetic effects. The investigators therefore undertook the present study to investigate whether preoperative dexamethasone could improve surgical outcome in patients undergoing thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thyroid surgery

Exclusion Criteria:

* ASA physical class III or IV
* age > 75 years
* pregnancy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing thyroid surgery for benign and malignant thyroidal disease
Sampling Method: Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela M CECILIA, M.D., Principal Investigator — Università degli Studi dell'Aquila
Locations (1):
- ospedale San Salvatore-Reparto di Chirurgia Generale Universitaria, L’Aquila, AQ, Italy

REFERENCES:
- [Derived] Schietroma M, Cecilia EM, Carlei F, Sista F, De Santis G, Lancione L, Amicucci G. Dexamethasone for the prevention of recurrent laryngeal nerve palsy and other complications after thyroid surgery: a randomized double-blind placebo-controlled trial. JAMA Otolaryngol Head Neck Surg. 2013 May;139(5):471-8. doi: 10.1001/jamaoto.2013.2821. PMID 23681030 (Retraction: PMID 30325981 JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1089)